CLINICAL TRIAL: NCT04142073
Title: Advanced Wireless and Wearable Sensors for Patients With Critical Neonatal and Pediatric Congenital Heart Defects
Brief Title: CCU Wireless Vital Signs Monitoring
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Stephanie Rangel, Director CTU, Northwestern University
Other Study IDs: SX08072018
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: CCU Inpatients
Keywords: wireless vitals; vitals monitor; cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children under 18 years of age

SUMMARY:
This is a pilot study is to test a wireless, skin-sensor device against current technology in the CCU to monitor vitals

DETAILED DESCRIPTION:
This is a single center, prospective, observational study that will recruit subjects from Lurie Children's Hospital to test a wireless vitals monitor against the current vitals monitors used in the Cardiac Care Unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients under the age of eighteen admitted to the Lurie's Children's Cardiac Care Unit will be eligible to participate

Exclusion Criteria:

* Patients at imminent risk of death
* Patients with a skin abnormality that precludes assessment
* Patients with hyperbilirubinemia and requiring a need for UV light

Ages: 0 Months to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients under the age of eighteen admitted to the Lurie's Children's Cardiac Care Unit will be eligible to participate
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Percent agreement with pilot sensor and current standard of vital signs monitoring | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Rangel, Study Director — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States